CLINICAL TRIAL: NCT06900881
Title: Role of Kefir Mouth Wash in Oral Health Status Amelioration: An in Vivo Study
Brief Title: Role of Kefir Mouth Wash in Oral Health Status Amelioration
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, ZAHRAA HUSSEIN DAWOOD, Master's Student in Dentistry, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUPRVOO15
Record Dates: First submitted 2025-03-09; First posted 2025-03-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Plaque Induced Gingivitis; Halitosis; Oral Disease
Keywords: Kefir; Moderate gingivitis; Halitosis; Plaque; Oral Health Status
MeSH Terms: conditions — Halitosis; Mouth Diseases; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Upon verifying a diagnosis of moderate gingivitis, sixty individuals age 18 -28 years will be randomly allocated into two parallel groups each group will received a similar number of participant (n=30) with a1:1 allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Upon verifying a diagnosis of moderate gingivitis, sixty individuals will be randomly allocated into two parallel groups using the Research Randomizer program (v. 2.0, https://www.randomizer.org),to mitigate bias.
  This procedure will be managed by a practiced dentist who is not participating in the trial and is securely maintain under his exclusive control.
  Both mouthwashes will be contained in bottles of similar color and form, labeled with codes (A, B) to ensure experimental blinding. This blinding technique guaranteed that neither the participants nor the examiner and no data analyses aware of the specific mouthwash included in each bottle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Kefir Mouth Wash (Active Comparator): The experimental group will take 60 mL of kefir mouthwash (Yogourmet, France) which contains live probiotic strains and active bacterial and yeast cultures, including (Lactococcus lactis, Lactococcus cremoris, Lactococcus diacetylactis, Lactobacillus acidophilus, Saccharomyces cerevisiae, and Kluyveromyces lactis, and maltodextrin)mixed with milk with 3 percent fat (Pegah, Iran) .The milk will be heated to boiling point and then allow to cool to room temperature (25°C). After cooling, the kefir powder will be dissolved and culture for 24 hours, use 60 ml daily, split into 30 mL in the morning and 30 mL in the evening. To guarantee uniformity in the intervention, participants follow a set rinse technique.
  Participants will be instructed to use the respective mouthwash (Kefir mouth wash) twice daily for 1 minute, 30 minutes after brushing their teeth, after the mouthwash application, participants will be advised not to eat or drink anything for one hour to ensure accurate results.
  Interventions: Combination Product: Kefir Mouth Wash
- Chlorhexidine 0,12% Bio fresh Mouth Wash (Other): The control group will take 30 mL of 0.12% chlorhexidine Bio fresh mouthwash (Scirto Co for Bio fresh LIC)daily, split into 15 mL in the morning and 15 mL in the evening. To guarantee uniformity in the intervention, participants follow a set rinse technique.
  Participants will be instructed to use the respective mouthwash (chlorhexidine) for 28 days twice daily for 1 minute, 30 minutes after brushing their teeth, after the mouthwash application, participants will be advised not to eat or drink anything for one hour to ensure accurate results.
  Interventions: Drug: Chlorhexidine 0,12%Biofresh Mouthwash

INTERVENTIONS:
Combination Product: Kefir Mouth Wash — A kefir-based mouthwash was developed with active bacterial and yeast cultures, including Lactococcus lactis, Lactococcus cremoris, Lactococcus diacetylactis, Lactobacillus acidophilus, Saccharomyces cerevisiae, and Kluyveromyces lactis, along with maltodextrin and 3% fat milk. The recipe also calls for milk from Pegah, Iran. The milk is initially heated to boiling point and then allowed to cool to room temperature (25°C). After cooling, the kefir powder will be dissolved in the cooled milk and mixed well. For every 1 liter of milk, 3g of kefir starter yogurt (Yogourmet, France) will be added. The inoculated milk will then be transferred into a clean, airtight container, and the lid will be sealed. The container will be left at room temperature for approximately 24 hours until the kefir curd forms. After 24 hours, the kefir will be refrigerated for about 8 hours to halt the fermentation process.
  Arms: Kefir Mouth Wash
Drug: Chlorhexidine 0,12%Biofresh Mouthwash — Chlorhexidine mouthwash is used as a standard treatment (Scitra Co for Biofresh LIC, P.O. Box 87218, Dubai, U.A.E.). It contains 0.12% Chlorhexidine Digluconate, purified water, sodium saccharin, cremophor, flavor, and glycerin.
  Arms: Chlorhexidine 0,12% Bio fresh Mouth Wash

SUMMARY:
The present research aims to evaluate the efficiency of kefir mouthwash in enhancing oral health status by employing an in vivo experimental approach. Specifically, the study will assess how kefir mouthwash influences key oral health indicators, including gingival inflammation, plaque development, oral hygiene status, and halitosis. The study will be conducted over a 28-day period, with follow-up assessments every 14 days. The study will include systemically healthy adults with moderate gingivitis. Clinical parameters such as the Gingival Index (GI), Plaque Index (PI), and Simplified Oral Hygiene Index (OHI-S) will be measured, along with inflammatory biomarkers, including Interleukin-1β (IL-1β) and Interleukin-10 (IL-10). Halitosis will be evaluated using a Hali meter device. All of these will be measured at base line and day 14 and day 28 end of the study. Chlorhexidine 0.12% will be used as a comparative control to evaluate the efficacy of kefir mouthwash in improving oral health. This research intends to provide scientific evidence supporting the use of kefir as a probiotic-based mouthwash, offering a natural alternative to chemical mouthwashes and potentially reducing the negative consequences commonly associated with their use.

DETAILED DESCRIPTION:
Due to their antibacterial qualities, conventional oral hygiene products such as chlorhexidine mouthwashes have been extensively used. However, their prolonged usage is often linked to negative effects, including taste changes, tooth discoloration, and mucosal discomfort. In response, natural and probiotic-based substitutes that provide efficient antibacterial activity with minimal adverse effects have attracted increasing attention. One such alternative gaining interest is kefir, a fermented milk product rich in antimicrobial peptides, probiotics, and bioactive components, which will be used in this study to assess the impact of kefir mouthwash on oral health.

The study will involve 60 systemically healthy adults aged 18 to 28 years, with moderate gingivitis. Participants will be selected from dental students at Bilad Al-Rafi Dain University and trained dentists from a specialist dental center in Diyala city. A triple-blind design will be used to eliminate bias, where the participants, the researchers administering the intervention, and the data analysts will all be blind to group assignments. Participants will be randomly assigned to one of two groups: the chlorhexidine 0.12% Bio Fresh group (Scirto Co for Bio Fresh LIC, P.O. Box 87218, Dubai, U.A.E.) or the kefir group (Yogourmet, France).

The research will span 28 days, with three data collection periods: baseline (Day 0), Week 2 (Day 14), and Week 4 (Day 28). Participants will use either kefir mouthwash or chlorhexidine 0.12% Bio Fresh mouthwash twice daily for one minute, 30 minutes after brushing their teeth, while refraining from eating or drinking for one hour after use. Both groups will receive mouthwashes in bottles that are identical in color and shape, labeled with random codes (A or B) to maintain blinding.

The chlorhexidine 0.12% Bio Fresh mouthwash will contain 0.12% Chlorhexidine Digluconate, purified water, sodium saccharin, Cremophor, flavoring, and glycerin, while the kefir mouthwash will be made using kefir powder containing live probiotic strains and active bacterial and yeast cultures, including Lactococcus lactis, Lactococcus cremoris, Lactococcus diacetylactis, Lactobacillus acidophilus, Saccharomyces cerevisiae, Kluyveromyces lactis, and maltodextrin, along with 3% fat milk.

The effectiveness of the mouthwashes will be assessed by evaluating the Plaque Index, Gingival Index, Simplified Oral Hygiene Index, and inflammatory cytokines (IL-1β and IL-10) at baseline, 14 days, and 28 days. Saliva samples will be collected at each follow-up to analyze the inflammatory response, and halitosis will be measured using the Hali Meter device. Participants will be monitored for compliance via daily tracking logs, electronic reminders through a WhatsApp group, and follow-up visits. Non-compliance or failure to adhere to the protocol will result in exclusion from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-28 years.
* Systemically healthy people without a history of chronic illness.
* Those suffering with moderate gingivitis.
* Not using any antibiotics over three months

Exclusion Criteria:

* History of systemic diseases.
* Pregnant, lactating females.
* History of antibiotic therapy in the past 3 months.
* History of oral prophylaxis within the last 6 months prior to the study as this can confound the results, making it difficult to determine the real effect of the mouthwash.
* Subjects with mouth breathing habits.
* Subjects with orthodontic and prosthodontic appliances.
* Subjects with deleterious habits such as smoking, because it may affect oral health status, causing periodontal disease, altered oral microbiota, and impaired healing. This can confound the study results, making it difficult to observe the mouthwash effect .
* Failure to follow the prescription regimen.
* Failure to follow the research protocol.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Changes in the clinical periodontal parameters of Gingival index | 0,14 ,28 days
  Gingival Index (GI):
  Subjects will undergo the measurement of the Gingival Index (GI), designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed based on color, consistency, and bleeding on probing. The unit of measurement for the Gingival Index (GI) is a numerical scale from 0 to 3, where each number represents the severity of gingival inflammation. Data will be collected based on the following four possible clinical conditions:
  Score 0 : Normal gingiva -no inflammation, healthy gums. Score1 : Mild Inflammation -slight change in color, slight edema, no bleeding on probing.
  Score 2 : Moderate Inflammation- redness, edema, and glazing; bleeding on probing.
  Score 3 : Severe Inflammation -marked redness and edema, ulceration, with a tendency for spontaneous bleeding.
Changes in clinical periodontal parameters of Plaque index | 0,14 ,28 days
  Plaque Index (PI):
  To determine the Plaque Index (PI) for participant, their dental plaque thickness is evaluated by probing the mesial, distal, buccal, and palatal surfaces of the teeth. During this evaluation, the probe is used to examine the presence of plaque. The individual plaque index will be determined by summing the values obtained for each tooth and calculating the average.
  scale as unit of measurement. The scoring system for the Plaque Index (PI) is as follows:
  Score 0 : No plaque-no plaque is present on any of the surfaces being probed. Score1 : Slight plaque- a small amount of plaque is visible at the gingival margin (border of the gum), but it is not abundant.
  Score2 : Moderate plaque- plaque is visible in moderate amounts, covering a larger portion of the tooth surface.
  Score 3 : Abundant plaque- a significant amount of plaque is present, covering most or all of the tooth surface.
Assessment of Oral Hygiene Status Using the Simplified Oral Hygiene Index | 0,14 ,28 days
  The Simplified Oral Hygiene Index (SOHI) is used to assess the oral hygiene status of participants by evaluating the amount of plaque and calculus present on their teeth. Using scale 0-3 as unit of measurement.
  The scoring system is as follows:
  Score 0 : Excellent Oral Hygiene- no plaque or calculus is present on the teeth.
  Score 1 : Good Oral Hygiene-small amounts of plaque or calculus are present, but they do not significantly affect oral health.
  Score 2 :Fair Oral Hygiene- moderate plaque or calculus accumulation is observed, indicating a need for improvement in oral hygiene practices.
  Score 3 : Poor Oral Hygiene-heavy plaque and/or calculus buildup is present, indicating poor oral hygiene practices and a need for immediate intervention.
  In this assessment, participants are evaluated based on these categories, with lower scores representing better oral hygiene and higher scores indicating a worse hygienic state.
Changes in the level of Halitosis | 0,14 ,28 days
  The Hali Meter Device (YRY Smart Breath Odor Detector) will be used to measure oral malodor (halitosis) by identifying volatile sulfur compounds (VSCs) . The severity of halitosis will be categorized into four levels based on the social distance cm at which the odor is detectable:
  Level 1 (Green light): Slight odor (20-65 cm)
  Level 2 (Yellow light): Moderate odor (65-90 cm)
  Level 3 (Pink light): Strong odor (90-120 cm)
  Level 4 (Red light): Intense odor (>120 cm)
  Measurement Method:
  Preparation: Subjects would refrain from eating, drinking, or performing oral hygiene for at least 1 hour before measurement .
  Test Initiation: The test would begin when the device vibrates and a blue light flashes.
  Measurement: The subject would blow into the device for 5 seconds, 1 cm away, and the corresponding light color would indicate the severity of halitosis. The results would be saved after pressing the top of the device.

SECONDARY OUTCOMES:
Changes in the level of inflammatory cytokines IL-1β by unstimulated saliva collection | 0,14 ,28 days
  2 mL of unstimulated saliva will be collected from all participants at baseline, and after 14 and 28 days, to measure changes in inflammatory cytokines IL-1β using the Enzyme-Linked Immunosorbent Assay ELISA technique.
  Unit of measurement . pg/L picograms per Liter as unit of measurement for IL-1β .
Changes in the level of inflammatory cytokines IL10 by unstimulated saliva collection | 0,14 ,28 days
  2 mL of unstimulated saliva will be collected from all participants at baseline, and after 14 and 28 days, to measure changes in inflammatory cytokines IL-10 using the Enzyme-Linked Immunosorbent Assay ELISA technique.
  Unit of measurement:
  ng/ml nanogram per milliliter as unit of measurement for IL10.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra H Al-Tamimi, MS student, Principal Investigator — Department of prevention, College of dentistry , University of Mustansiriyah
Locations (1):
- Al-Mustansiriyah University/College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No